CLINICAL TRIAL: NCT02489656
Title: Effect of a Silicone Hydrocoated Double Loop Ureteral Stent on Symptoms and Quality of Life in Patients Undergoing F-URS for Kidney Stone; a Comparative Randomized Multicenter Clinical Study.
Brief Title: Quality of Life in Patients With Double Loop Ureteral Stent (JJ Silicone Hydrogel Study)
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Coloplast A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DUDLUIV1201EC
Record Dates: First submitted 2015-05-18; First posted 2015-07-03 (Estimated); Last update posted 2015-07-03 (Estimated); Status verified 2015-05

CONDITIONS: Kidney Calculi
Keywords: Double loop ureteral stent; USSQ; Quality of life; Pain
MeSH Terms: conditions — Kidney Calculi; Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Coloplast Hydrocoated silicone JJ stent (Experimental): Double loop ureteral stent endoscopic placement
  Interventions: Device: Double Loop Ureteral stent endoscopic placement.
- Boston Percuflex Plus JJ stent (Active Comparator): Double loop ureteral stent endoscopic placement
  Interventions: Device: Double Loop Ureteral stent endoscopic placement.

INTERVENTIONS:
Device: Double Loop Ureteral stent endoscopic placement. — A JJ stent placement may be indicated at the end of the endourological removal of kidney stones to ensure urine drainage and cicatrisation

SUMMARY:
This study is a prospective, randomized multicenter study conducted in Europe. It is designed to compare two double loop ureteral stents in terms of the quality of life in patients operated on a kidney stone and requiring the placement of a double loop ureteral stent at the end of the operation.

DETAILED DESCRIPTION:
* The double loop stents are used for both prevention and treatment of ureteral obstruction: They permit the interim internal bypass drainage of urine when obstruction in the ureter especially in cases of lithiasis or after surgical intervention on the upper urinary tract.
* There are many indications for double loop stent placement and population chosen for this study are adult patients with intra-renal calcium calculi of 7-20 mm in diameter for whom the treatment indication is a flexible ureterorenoscopy.
* The aims of the use of a double loop stent are to

  * prevent complications (pain, infection) associated with the ureteral obstruction by any residual stone fragments, blood clot or local oedema generated by the intervention.
  * preserve the renal function.
  * facilitate healing process while limiting the risk of stenosis and probably reduce the rate of readmission after patients' discharge.
* Double loop Stent-related symptoms have a high prevalence and may affect over 80% of patients.
* Assessment tools are important to determine the symptoms intensity and allow for comparisons at different times. The Urinary Stent Symptom Questionnaire (USSQ) is the most adapted tool designed for this purpose.
* An ideal ureteral stent is expected to drain well, to be easy to insert and to be comfortable for the patients. The investigators designed a hydro-coated Silicone JJ stent with additional properties for improving patient's comfort.
* The investigators decided to perform a randomized clinical investigation to evaluate the Coloplast Hydrocoated Silicone JJ in comparison to the Boston Percuflex Plus JJ stent on patients' comfort.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female patients
2. Aged > 18 years
3. Unilateral renal non-infection stone for whom the treatment indication is a flexible ureterorenoscopy (multiple kidney stones are acceptable provided that only one side is currently symptomatic)
4. Index stone of 5-25 mm (measured on plain abdomen X-Ray KUB or CT)
5. Without any currently implanted JJ stent
6. Patient agreed to participate to the study and having signed the consent form
7. Able to complete self-rated questionnaires.

Exclusion Criteria:

1. Acute ureteric/nephritic colic (residual pain is acceptable)
2. Any type of chronic pain
3. Large stones > 25 mm
4. Infection renal stone already diagnosed and documented
5. Malformation of urinary tract (e.g. Horseshoe kidney, duplicity or, ureterocele, mega ureter)
6. Diverticulum stone
7. Urogenital tumor
8. Any significant neurological disease or injury impacting sensation
9. JJ stents already implanted
10. Patients with long-term indwelling urethral catheter
11. No indication for JJ insertion (e.g. spontaneous stone passage)
12. Untreated urinary tract infection
13. Ureteral obstruction (stenosis, compression, calculi)
14. Neurogenic bladder
15. Overactive bladder
16. Bladder stone
17. Chronic prostatitis
18. BPH treated (recent initiation of 5 alpha-Reductase Inhibitor or Phytotherapeutic agents)
19. Ongoing Alpha-Blocker or Anticholinergic medication
20. Pregnancy
21. Any event discovered during the endoscopy which is not compatible with the study design and objective

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2013-09; Primary Completion 2016-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
USSQ scale (Ureteral Stent Symptoms Questionnaire) | at day 20

SECONDARY OUTCOMES:
Evaluate impact on quality of life via the USSQ questionnaire assessing 5 other scores and adverse event reporting at all visits. | Day 2, 7 and 35

OTHER OUTCOMES:
Encrustation of double loop ureteral stents | after 20 days (JJ stent removal)
  Encrustation of double loop ureteral stents is evaluated by a score of integer values ranging from 0 to 6

CONTACTS AND LOCATIONS:
Overall Officials: Olivier PJ Traxer, Professor, Principal Investigator — Service de Chirurgie Urologique de l'Hôpital Tenon
Locations (1):
- Service de Chirurgie Urologique de l'Hôpital Tenon, Paris, France